CLINICAL TRIAL: NCT01728870
Title: Comparison of Partial Enteral Nutririon (Modulen) With a Unique Diet to Exclusive Enteral Nutrition (Modulen) for the Treatment of Pediatric Crohn's Disease. A Prospective Randomized Controlled Trial.
Brief Title: Partial Enteral Nutrition With a Unique Diet vs. Exclusive Enteral Nutrition for the Treatment of Pediatric Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Arie Levine (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Arie Levine, Director, Pediatric Gastroenterology and Nutrition unit., Wolfson Medical Center
Organization: Wolfson Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0164-12-WOMC
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Crohn's Disease
Keywords: Pediatric; Crohn's disease; Mild to moderate Crohn's Disease; Diet; Enteral Nutrition
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unique Diet+Partial Enteral Nutrition (Experimental): Unique Diet+Partial Enteral Nutrition (PEN): This group will receive as follows:
  Weeks 1-6: 50% of dietary needs from PEN (Modulen, Nestle) and 50% from a limited whole food diet.
  Weeks 7-12: 25% of dietary needs from PEN (Modulen, Nestle) and 75% from a limited whole food diet.
  Interventions: Other: Unique Diet+Partial Enteral Nutrition
- Exclusive Enteral Nutrition (Modulen) (Active Comparator): Exclusive Enteral Nutrition(EEN): This group will receive as follows:
  Weeks 1-6: EEN(100% of dietary needs from Modulen) Weeks 7-12: 25% of dietary needs from Modulen and 75% from a free diet.
  Interventions: Other: Exclusive Enteral Nutrition (Modulen)

INTERVENTIONS:
Other: Unique Diet+Partial Enteral Nutrition — Modulen - liquid dietary formula
  Other Names: Modulen, Nestle
  Arms: Unique Diet+Partial Enteral Nutrition
Other: Exclusive Enteral Nutrition (Modulen)
  Other Names: Modulen, Nestle
  Arms: Exclusive Enteral Nutrition (Modulen)

SUMMARY:
The purpose of this study is to assess the efficacy and tolerability of a novel dietary intervention for early CD based on partial enteral nutrition, and to compare it to the gold standard but difficult to implement dietary intervention- Exclusive enteral nutrition with Modulen .

DETAILED DESCRIPTION:
Background: Crohn's disease is clearly on the rise in countries exposed to industrialization and western diet. Several factors may implicate diet in the pathogenesis of CD or in disease activity. The strongest argument for an effect of diet is the effect of exclusive enteral nutrition (EEN) on disease activity in CD. 40-80% of children , fed an exclusive liquid diet, irrespective of which diet, will enter complete remission, often with normalization of inflammatory markers. The effect of formula has been shown to be independent of fat or protein composition in pediatric studies, but to be dependent on exclusion of normal diet.Thus, rather than the composition of EEN being associated with remission of disease it may be the exclusion of certain components of the Western diet may be responsible for improvement.

Methods:This is a prospective randomized controlled trial, in patients with a recent diagnosis of CD (up to two years),aged 4-18, comparing two arms over 12 weeks of therapy.

Group 1:will receive 50% of their dietary needs from a polymeric formula ( Modulen, Nestle) and a limited whole food diet for 6 weeks/ Group 2: will receive EEN with Modulen for 6 weeks. At the end of 6 weeks, all patients entering remission (irrespective of randomization) will enter the second 6 week phase, continuing 25 % of calories as Modulen in both groups. Patients in remission from group 2 will continue to consume 25% of calories as Modulen and be allowed free diet , patients in Group 1 will continue 25% of calories from Modulen but continue restricted diet.

Patients will be seen at onset (week 0), weeks 3 and 6, 12 and 24 weeks.

We hypothesize that by withdrawing the offending dietary agents we can achieve an equal remission rate with improved tolerability. This study will evaluate response, remission and tolerability in both groups, as well as the effects of nutrition on bone health.

ELIGIBILITY:
Inclusion Criteria:

1. Children 4-18 years of age.
2. Patients with a diagnosis of CD-duration of disease up to 36 months
3. Have macroscopic small bowel involvement, or isolated large bowel disease confined to the right or transverse colon
4. Patients with a pediatric activity index -PCDAI ≥ 10
5. Patients will not be excluded if they have received 5ASA or an immunomodulator for >8 weeks and the dose is stable , or if they start a thiopurine concurrently , as thiopurines are not considered sufficient to induce remission in active disease before 8 weeks as an isolated therapy.
6. Informed Consent

Exclusion Criteria:

1. Patients with no disease activity ( PCDAI <10) or severe disease ( PCDAI ≥ 40).
2. Patients who have received corticosteroids of any kind in the previous 4 weeks.
3. Patients who have started an immunomodulator in the previous 8 weeks
4. Any current biological treatment
5. Isolated Large bowel disease ( L2) involving the recto-sigmoid or descending colon
6. Patients with penetrating disease (abscess or fistula)
7. Active Perianal disease
8. Fixed stricture or small bowel obstruction
9. Normal CRP and ESR
10. Active joint disease.
11. Patients who have undergone an intestinal resection.
12. Sclerosing Cholangitis
13. Pregnancy

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2013-01; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
patient's adherence with the diet assessed by cessation of therapy because of patients refusal to continue and by a MARS questionnaire | 6 weeks

SECONDARY OUTCOMES:
Response, defined as a drop in PCDAI of 12.5 points or remission, on an intention to treat analysis. | 6 weeks
Remission at week 6 and week 12 (defined as PCDAI≤10, or less than 7.5 without height component), | 6 weeks and 12 weeks
Bone health | at the 3, and 6 month visits
  change in serum bone biomarkers from baseline and their correlation with DEXA (optional)
CRP at week 12 | 12 weeks
Physician assessment of compliance | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arie Levine, MD, Principal Investigator — Pediatric Gastroenterology and Nutrition unit, Wolfson MC
Locations (3):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - IWK Health Centre, Halifax, Nova Scotia
- The E. Wolfson.Medical Center, Holon, Israel

REFERENCES:
- [Derived] Sigall Boneh R, van der Kruk N, Wine E, Verburgt CM, de Meij TGJ, Lowenberg M, Gecse KB, Wierdsma N, Derikx JPM, de Jonge WJ, D'Haens G, Ghiboub M, Van Limbergen JE. Tryptophan metabolites profile predict remission with dietary therapy in pediatric Crohn's disease. Therap Adv Gastroenterol. 2025 Feb 25;18:17562848251323004. doi: 10.1177/17562848251323004. eCollection 2025. PMID 40012837
- [Derived] Verburgt CM, Dunn KA, Ghiboub M, Lewis JD, Wine E, Sigall Boneh R, Gerasimidis K, Shamir R, Penny S, Pinto DM, Cohen A, Bjorndahl P, Svolos V, Bielawski JP, Benninga MA, de Jonge WJ, Van Limbergen JE. Successful Dietary Therapy in Paediatric Crohn's Disease is Associated with Shifts in Bacterial Dysbiosis and Inflammatory Metabotype Towards Healthy Controls. J Crohns Colitis. 2023 Jan 27;17(1):61-72. doi: 10.1093/ecco-jcc/jjac105. PMID 36106847
- [Derived] Ghiboub M, Penny S, Verburgt CM, Boneh RS, Wine E, Cohen A, Dunn KA, Pinto DM, Benninga MA, de Jonge WJ, Levine A, Van Limbergen JE. Metabolome Changes With Diet-Induced Remission in Pediatric Crohn's Disease. Gastroenterology. 2022 Oct;163(4):922-936.e15. doi: 10.1053/j.gastro.2022.05.050. Epub 2022 Jun 7. PMID 35679949
- [Derived] Sigall Boneh R, Van Limbergen J, Wine E, Assa A, Shaoul R, Milman P, Cohen S, Kori M, Peleg S, On A, Shamaly H, Abramas L, Levine A. Dietary Therapies Induce Rapid Response and Remission in Pediatric Patients With Active Crohn's Disease. Clin Gastroenterol Hepatol. 2021 Apr;19(4):752-759. doi: 10.1016/j.cgh.2020.04.006. Epub 2020 Apr 14. PMID 32302709
- [Derived] Levine A, Wine E, Assa A, Sigall Boneh R, Shaoul R, Kori M, Cohen S, Peleg S, Shamaly H, On A, Millman P, Abramas L, Ziv-Baran T, Grant S, Abitbol G, Dunn KA, Bielawski JP, Van Limbergen J. Crohn's Disease Exclusion Diet Plus Partial Enteral Nutrition Induces Sustained Remission in a Randomized Controlled Trial. Gastroenterology. 2019 Aug;157(2):440-450.e8. doi: 10.1053/j.gastro.2019.04.021. Epub 2019 Jun 4. PMID 31170412